CLINICAL TRIAL: NCT04023643
Title: Pragmatic And Randomized Pediatric Ventilation Weaning Trial
Brief Title: Pediatric Ventilation Weaning
Acronym: PROVENTUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: São Paulo State University (Other)
Collaborators: Andréa Maria Cordeiro Ventura (Unknown)
Responsible Party: Principal Investigator, Murilo Lourenção, Principal investigator, São Paulo State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90326618.7.1001.0076
Record Dates: First submitted 2019-07-12; First posted 2019-07-17 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Respiration, Artificial; Ventilator Weaning
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP + PS (Experimental): Weaning from mechanical ventilation using CPAP + PS
  Interventions: Other: Ventilation Weaning
- SIMV + PS (Active Comparator): Weaning from mechanical ventilation using SIMV+PS
  Interventions: Other: Ventilation Weaning

INTERVENTIONS:
Other: Ventilation Weaning — Use of different weaning strategies

SUMMARY:
The hypothesis of the present study is that the use of Continuous Positive Airway Pressure (CPAP) plus PS can accelerate the weaning process and, consequently, shorten the MV. This multicenter, pragmatic clinical trial aims to compare the use of CPAP + PS versus SIMV + PS as a method for ventilatory weaning of children, emphasizing the duration of the process. There are no similar studies in the world.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) is a widely used practice among Pediatric Intensive Care Units (PICUs) throughout the world. Data from multicenter studies reveal rates ranging from 20% to 64% use, lasting about 5 to 6 days.

The practice of using artificial methods to provide respiratory care is considered a revolution in the care of critically ill patients, reducing their morbidity and mortality. On the other hand, it is widely known that these tools bring with it a myriad of possible complications, such as Health Care-Associated Pneumonia, upper and lower airway injuries, risks related to sedation, and cardiovascular instability. Therefore, it is indispensable to interrupt the MV as soon as possible.

When is spent a lot of time recognizing that the MV is no longer essential, is increased the risks and costs (up to $ 2,000 a day), and is failed the good medical practice. Currently, the duration of weaning consumes about 40% of the total MV time. This depends on many factors, such as fluid balance, positive end expiratory pressure (PEEP), sedation, pulmonary hypertension and diaphragm function, among others.

Studies have shown that the implementation of a weaning protocol reduces its duration and, consequently, ventilation in children. There are numerous known weaning techniques, however, the most commonly used approach is the progressive reduction of ventilatory support already in use, maintaining the same modes and reducing the parameters. Some professionals choose synchronized intermittent mandatory ventilation (SIMV), reducing respiratory rate, with or without Supplementary Pressure (PS) association. Others prefer to perform daily extubation readiness tests (ERT) or to switch spontaneous breathing methods with full-support ventilation for respiratory muscle training, this practice is more common in adult ICUs. Exhorted by recommendations for mechanical ventilation of critically ill children at the 2017 pediatric mechanical ventilation consensus conference (PEMVECC), who concluded with strong agreement that there is insufficient data to recommend the method for weaning the investigators decided to study the assertive.

ELIGIBILITY:
Inclusion Criteria:

* Children who underwent mechanical ventilation for at least 24 hours in one of the participant PICUs

Exclusion Criteria:

* Children dependent on mechanical ventilation and / or chronically supplemental oxygen;
* Children with do not resuscitation order (DNR)
* Children with neurological and neuromuscular disorders that may interfere with MV;
* Children with chronic lung diseases (such as cystic fibrosis, bronchopulmonary dysplasia, chronic obstructive pulmonary disease, with the exception of asthma);
* Children transferred from another PICU not included in the trial and whose weaning has already begun;
* Children whose cannulae have air leakage higher of 25% of inspiratory flow, without indication for cannula replacement.

Ages: 29 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Ventilator-free days | 4 days
  Rate of free days of mechanical ventilation during ICU admission in children who were intubated. Assessed by the data collection form filled daily by the collaborators.
Rate of Weaning duration | 12 hours
  Amount of hours spent in ventilator weaning. Assessed by the data collection form filled daily by the collaborators.

SECONDARY OUTCOMES:
Rate of PICU length of Stay | 10 days
  Amount of days spent in PICU. Assessed by the data collection form filled daily by the collaborators.
Incidence of Complications associated with mechanical ventilation | 10 days
  Incidence of Health Care associated Pneumonia; tracheitis; barotrauma; extubation laryngitis. Diagnosed according to the protocols in force at the institution and Assessed by the data collection form filled daily by the collaborators.
Rates of spontaneous breathing test failure | 6 days
  Rates of spontaneous breathing test failure. Assessed by the data collection form filled daily by the collaborators.

CONTACTS AND LOCATIONS:
Overall Officials: Murilo Lourenção, MD, Principal Investigator — HU-USP; Andrea Ventura, MSC, MD, Study Director — HU-USP
Locations (5):
- Brazil (5):
  - Hospital das Clínicas de Marília - Unidade II, Marília, São Paulo
  - Hospital Municipal Vila Santa Catarina, São Paulo
  - Hospital Municipal Dr. Moysés Deutsch, São Paulo
  - Instituto da Criança do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
  - Hospital Universitário da Universidade de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR